CLINICAL TRIAL: NCT05416658
Title: Examining the Effectiveness of a Shared Decision Making Intervention for Antipsychotic Medications to Improve Engagement in Treatment for People Experiencing Early Psychosis
Brief Title: Shared Decision Making for Antipsychotic Medications
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: New York State Psychiatric Institute (Other)
Collaborators: Temple University (Other)
Responsible Party: Principal Investigator, Lisa Dixon, Edna L. Edison Professor of Psychiatry, New York State Psychiatric Institute
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: 1R34MH128497-01A1 (NIH)
Record Dates: First submitted 2022-06-03; First posted 2022-06-13 (Actual); Last update posted 2025-03-20 (Actual); Status verified 2025-03

CONDITIONS: Schizophrenia; Schizoaffective Disorder; Schizophreniform Disorders; Delusional Disorder; Other Specified Schizophrenia Spectrum and Other Psychotic Disorder
Keywords: Shared decision making; psychosis; schizophrenia; antipsychotic; medication; intervention; decision aid; coordinated specialty care (CSC); randomized controlled trial (RCT)
MeSH Terms: conditions — Schizophrenia; Psychotic Disorders; Schizophrenia, Paranoid

STUDY DESIGN:
Who Masked: Care Provider
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- The Antipsychotic Medication Decision Aid (APM-DA) intervention clinics (Experimental): Three pairs of comparable clinics (out of 22 clinics where OnTrackNY operates) based on the same region of the state and similar numbers of patients with similar demographic composition. One of each paired clinic is assigned to the intervention group by a blinded Co-I who will generate binary random variables.
  Interventions: Other: The Antipsychotic Medication Decision Aid (APM-DA)
- Treatment As Usual (TAU) clinics (No Intervention): The other clinic of each of the three pairs will be assigned to TAU.

INTERVENTIONS:
Other: The Antipsychotic Medication Decision Aid (APM-DA) — The APM-DA intervention is the first and only International Patient Decision Aid Standards (IPDAS) approved shared decision making (SDM) decision aid intervention for Antipsychotic Medication decisions in psychiatric visits. The APM-DA intervention developed by the research team addresses a common issue among psychiatric care providers and patients that lies in the heart of pharmacotherapy - taking, tapering or stopping APM. The APM-DA has a print format and can be used online as a PDF. It includes a concise table describing what each option involves, its benefits, risks, and strategies to reduce risks. The intervention was developed in co-production with various stakeholders (patients, clinicians, service leadership, family members, researchers). Additional intervention materials are an evidence document to support the information and an APM side effects table.
  Arms: The Antipsychotic Medication Decision Aid (APM-DA) intervention clinics

SUMMARY:
This study aims to provide an evidence-based shared decision making intervention for antipsychotic medications, the Antipsychotic Medication Decision Aid (APM-DA), for individuals experiencing early psychosis and provide, for the first time, an understanding of the shared decision making mechanism of action.

DETAILED DESCRIPTION:
The investigators will conduct a cluster RCT of the APM-DA intervention at 6 OnTrackNY clinics, with 3 clinics implementing APM-DA as part of their psychiatric visits and 3 randomized to serve as control offering treatment as usual (TAU). The planned sample size is 120 OnTrackNY clients with first episode psychosis (FEP). This real-world pilot cluster RCT will assess the feasibility of the APM-DA intervention in FEP care, providing the first evidence for the effectiveness of the APM-DA compared with TAU and understanding of the SDM intervention's mechanism of action.

ELIGIBILITY:
Inclusion Criteria:

* Ages 18 to 30 who have experienced nonaffective psychosis with a diagnosis of schizophrenia, schizoaffective disorder, schizophreniform disorder, delusional disorder, other specified/unspecified schizophrenia spectrum and other psychotic disorders (ICD-10-CM Diagnosis Code F20.x)
* Current/past experiences with antipsychotic medications (APM; e.g., currently taking any antipsychotic medication, stopped taking, or considering stopping).
* Receive FEP treatment in one of OnTrackNY clinics/sites randomized to intervention or treatment as usual (TAU) - Willing to participate in research interviews after each APM visit during the study period (3 months)

Exclusion Criteria:

* Unable to provide informed consent
* No experience with APM
* Not fluent (speaking, reading, writing) in English

Ages: 18 Years to 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 120 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2026-06-30 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
The 9-item Shared Decision Making Questionnaire for Psychiatry (SDM-Q-9-Psy) (Primary) | Change in SDM from baseline (T0, measured after the first medication visit) to the next post medication visit/s (Tnext) and up to a period of 3 months follow-up (T2)
  The 9-item Shared Decision Making Questionnaire for Psychiatry (SDM-Q-9-Psy) is the only validated self-report measure for SDM in psychiatry/mental health. The SDM-Q-9-Psy includes 9 items ranging from 0 to 5, with higher scores indicating higher quality of the SDM process perceived by the patient. The SDM-Q-9-Psy will be first measured (baseline, T0) after the first medication visit and then after each medication visit throughout the study period, therefore there will be multiple post-visits or "Tnext".
Intent to Attend and Complete Treatment Scale (Primary) | Change in OnTrackNY engagement from baseline (T0, measured at enrollment), after each post medication visit/s (Tnext), and at 3-month follow-up (T2 )
  The Intent to Attend and Complete Treatment are two items that are part of the EPINET Core Assessment Battery (CAB) "Medication Side Effects and Treatment Adherence" core domain to assess engagement in CSC program (OnTrackNY). The score ranges from 0 to 9 for each item, with higher scores indicating higher intent to attend and complete treatment. Changes in the Intent to Attend will be measured after each medication visit throughout the study period, therefore there will be multiple post-visits or "Tnext".
Adherence Estimator (Primary) | Change in Adherence Estimator from baseline (T0, measured at enrollment), after each post-visit/s (Tnext), and at 3-month follow-up (T2 )
  The Adherence Estimator is a three-item measure relies on client self-report. The Adherence Estimator focuses on perceived concerns about medications, perceived need for medications, and perceived affordability of medications. The Adherence Estimator is scored by adding up the total number of points in each item and can range from 0 (Low risk for adherence problems) to 36 (High risk for adherence problems). Changes in the Adherence Estimator will be measured after each medication visit throughout the study period, therefore there will be multiple post-visits or "Tnext".

IPD SHARING:
Plan to Share IPD: Yes
Findings from this study will be presented to research peers, clinicians, and the public through Presentations at Scientific Meetings, Regional Research or Educational Meetings, Newsletters and Social Media and Peer-Reviewed Publications. Those events will occur during or at the conclusion of the study.
Time Frame: Descriptive and raw data will be submitted on an annual basis. Unpublished de-identified data will be shared within one year after project completion, or when the data are published, whichever is earlier.
Access Criteria: Data and materials will be made available for research to investigators working under a Federal Wide Assurance who meet security measures and data use agreement criteria associated with public repositories, including the National Database for Clinical Trials related to Mental Illness (NDCT) and the NIMH Database of Cognitive Training and Remediation Studies (DoCTRS).